CLINICAL TRIAL: NCT00802061
Title: Sleep at 30 Degrees in Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: Trope 003
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Glaucoma
Keywords: progressive glaucoma despite controlled IOP
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Sleeping position in glaucoma patient

SUMMARY:
This study is designed to investigate the effect of body posture (particularly when sleeping) on the pressure in the eye. The effect of body posture on progressive glaucoma (glaucoma where a significant change i.e. a disc hemorrhage has occurred) is not known.

The study will involve being admitted to the Sleep Unit of the University Health Network at Toronto Western Hospital for 1 night (14 hours). IOP will be measured in both eyes every 2 hours with a Tonopen, along with brachial blood pressure (BP), in the sitting position until the patients reach their normal sleep cycle time. Patients will then be asked to sleep in either lying down or reclining at a 30 degrees position and have the IOP measurements and brachial BP every 2 hours in that position.

The same cohort of patients will then be invited for a repeat 14 hour IOP and BP measurement but will change their position, i.e. sitting before will now be supine and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* This pilot study included patients with progressive NTG or POAG as evidenced by disc hemorrhage despite well controlled Intraocular pressures (IOP), who were able to sleep flat

Exclusion Criteria:

* Any patients who were not able to sign a consent or lying flat during sleep

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada